CLINICAL TRIAL: NCT04982380
Title: Efficacy and Safety of Combined Bifidobacterium, Lactobacillus, Enterococcus and Bacillus Cereus Tablets, Live (Siliankang) in Patients With Type 2 Diabetes and Constipation: a Randomized, Double-blind, Placebo-controlled, Multicenter Trial
Brief Title: Efficacy and Safety of Bifidobacterium Quadruple Live Tablets in Patients With T2DM and Constipation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: First Affiliated Hospital of Harbin Medical University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Affiliated Hospital of Chengde Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Chinese Academy of Sciences (Other Government); Hangzhou Grand Biologic Pharmaceutical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLK-HS2843
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes Mellitus With Complication
Keywords: Type 2 diabetes;Constipation;Gut microbiota;Bifidobacterium
MeSH Terms: interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients will be instructed to continue current antidiabetic treatment, which should be kept unchanged throughout the trial, and start treatment with Bifidobacterium, Lactobacillus, Enterococcus and Bacillus Cereus Tablets, Live (Siliankang) 3 tablets p.o. tid for 12 weeks.
  Interventions: Drug: Bifidobacterium, Lactobacillus, Enterococcus and Bacillus Cereus Tablets, Live
- Control group (Placebo Comparator): Patients will be instructed to continue current antidiabetic treatment, which should be kept unchanged throughout the trial, and start treatment with Siliankang simulative tablets 3 tablets p.o. tid for 12 weeks.
  Interventions: Drug: Siliankang simulating tablets

INTERVENTIONS:
Drug: Bifidobacterium, Lactobacillus, Enterococcus and Bacillus Cereus Tablets, Live — Patients will be instructed to continue current antidiabetic treatment, which should be kept unchanged throughout the trial, and start treatment with Bifidobacterium, Lactobacillus, Enterococcus and Bacillus Cereus Tablets, Live (Siliankang) 3 tablets p.o. tid for 12 weeks.
  Other Names: Siliankang
  Arms: Experimental group
Drug: Siliankang simulating tablets — Patients will be instructed to continue current antidiabetic treatment, which should be kept unchanged throughout the trial, and start treatment with Siliankang simulative tablets 3 tablets p.o. tid for 12 weeks.
  Arms: Control group

SUMMARY:
Constipation is one of the common complication of diabetes mellitus, whose pathogenesis was previously recognized as decreased gastrointestinal motility caused by diabetic autonomic neuropathy. It is always treated with gastrointestinal motility drugs or laxatives which may have side effects such as gut microbiota dysbiosis and withdraw symptoms. Recently, researches have indicated that the risk of developing type 2 diabetes mellitus is associated with alterations in the structure of the gut microbiota and have begun to treat diabetic constipation by improving gut microbiota of these patients. The rational use of microecological preparation for the prevention and treatment of diabetic constipation has received increasing attention. This trial is aimed to evaluate the efficacy and safety of Combined Bifidobacterium, Lactobacillus, Enterococcus and Bacillus Cereus Tablets, Live (Siliankang) in the treatment of patients with type 2 diabetes and constipation, and to analyze its influence on gut microbiota and blood glucose.

DETAILED DESCRIPTION:
This is a 16 week, 1:1 randomised, controlled, open label, two-arm, parallel-group trial evaluating efficacy and safety of Combined Bifidobacterium, Lactobacillus, Enterococcus and Bacillus Cereus Tablets, Live (Siliankang) in patients with type 2 diabetes and constipation. Patients will be randomized into experimental group or control group treated with Siliankang or placebo tablets respectively. Total trial duration for the individual subject will be approximately 16 weeks including screening, 12-weeks treatment and 4-weeks follow-up. Patients will attend at 2-week, 8-week, 12-week and 16-week throughout the trial taking physical examination, having blood test, collecting faecal specimen and completing the questionnaire of constipation under the direction of doctors.

ELIGIBILITY:
Inclusion Criteria:

* According to the diagnostic criteria of World Health Organization (WHO) in 1999, type 2 diabetes mellitus was diagnosed clinically. The duration of T2DM was no more than 8 years (including 8 years).
* According to the ROME III diagnostic criteria of functional constipation or guideline for diagnosis and treatment of chronic constipation in China (2013 edition), chronic constipation was diagnosed clinically. The duration of constipation was more than 6 months (including 6 months).
* The age ranged from 18 to 70 years (including 18 and 70 years) with no restriction of sex.
* Fasting blood glucose was no more than 8mmol/L and glycosylated hemoglobin ranged from 7.0% to 10.0% (including 7.0% and 10.0%).
* Sign written consent form voluntarily.

Exclusion Criteria:

* Other types of diabetes mellitus.
* History of diabetic ketoacidosis and hyperosmolar hyperglycemic syndrome.
* Constipation induced by drugs[i.e. antidepressants, calcium antagonists, diuretics, sympathetic agents, antacids with aluminum or calcium, calcium agents, iron agents, antidiarrhetics].
* Organic constipation [i.e. intestinal diseases，endocrine and metabolic diseases (except diabetes), nervous system and muscle disease].
* Gastrointestinal diseases [i.e. colitis, mesenteric lymphadenitis, with a history of intestinal surgery].
* Using drugs that may affect clinical outcome evaluation in the past 2 weeks, such as antibiotics (penicillin, amoxicillin, erythromycin, azithromycin and cephalosporin, etc.), microecological preparations, laxative drugs (magnesium sulfate and lactulose, etc.); anthraquinones (rhubarb, aloe and senna, etc.); Gastrointestinal motility drugs (metoclopramide, domperidone, cisapride, etc).
* History of myocardial infarction or stroke within 6 months, or existing severe cardiovascular disease and risk.
* Abnormal liver function [i.e. serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is 1.5 times higher than the upper limit of normal value]. Abnormal renal function [Creatinine exceeds the upper limit of normal value].
* Severe hypertension that defined as systolic blood pressure ≥160 mmHg, diastolic blood pressure ≥90 mmHg with drug therapy, or hypotension (resting seat blood pressure < 90/50 mmHg).
* History of acute and chronic gastroenteritis or gastrointestinal surgery
* Psychosis, alcohol dependence or history of drug abuse.
* Lactating women, pregnant women and patients who have pregnancy plan during the trial or within 3 months after the trial.
* Participation in other studies three months before the trial.
* Allergic constitution or allergic to a variety of drugs.
* Those researchers think inappropriate to the research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-07-31 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of bowel movements | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  Changes from baseline in the number of completely spontaneous bowel movements (CSBMs) and number of spontaneous bowel movements (SBMs). Effectiveness is defined as CSBMs more than 3 times weekly (including 3 times) with increase from baseline, while ineffectiveness is defined as CSBMs less than 3 times weekly or with no increase from baseline.
Glycosylated hemoglobin | Baseline, Week 12, Week 16
  Changes from baseline in glycosylated hemoglobin.
Glycosylated albumin | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  Changes from baseline in glycosylated albumin.

SECONDARY OUTCOMES:
Gut micobiota | Baseline, Week 4, Week 8, Week 12, Week 16
  Changes from baseline in gut microbiota.
The ratio of CSBMs to SBMs | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  Changes from baseline in the ratio of CSBMs to SBMs.
Bristol Stool Scale | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  Proportions whose stool characters recover to Type III and IV by Bristol Stool Scale.
Bowel Function Index (BFI) | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  Changes from baseline in the score of Bowel Function Index (BFI).
Patient Assessment of Constipation symptom (PAC-SYM) | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  Changes from baseline in the scale of Patient Assessment of Constipation symptom (PAC-SYM).
Patient global impression of changes (PGIC) | Week 16
  Difference in the Patient global impression of changes (PGIC) between experimental group and control group.
The first time of CSBM | Week 1 to Week 16
  Difference in the first time of completely spontaneous bowel movement (CSBM) between the experimental group and control group.
Fasting blood glucose | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  Changes from baseline in fasting blood glucose.
Serum lipid spectrum | Baseline, Week 12
  Changes from baseline in serum lipid spectrum.

CONTACTS AND LOCATIONS:
Overall Officials: Weigang Zhao, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No